CLINICAL TRIAL: NCT03396237
Title: Vitamin D Deficiency Among Women With Unexplained Infertility
Acronym: Infertility
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Bahaa Eldin Ahmed, Clincal professor, Ain Shams Maternity Hospital
Other Study IDs: Vitamin D and Infertility
Record Dates: First submitted 2018-01-05; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Case Control Study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Case group contain cases of unexplained infertility women
- Group B: Control group contain fertile pregnant women

SUMMARY:
Does vitamin D is more deficient in women with unexplained infertility than in fertile pregnant women or not?

DETAILED DESCRIPTION:
The study will be done on women with unexplained infertility as a case group and fertile pregnant women as control group to detect if there's a difference in serum level of vitamin D between two groups which will help in the future for curing unexplained infertility women.

ELIGIBILITY:
Inclusion Criteria:

* women with unexplained infertility.
* pregnant fertile women as control group.

Exclusion Criteria:

* • Endocrinopathies such as (diabetes mellitus, thyroid disorders, parathyroid disorders and hyperprolactinemia), cardiovascular related diseases, severe infection, malignancies and concomitant diseases contribute to Vit D deficiency.

  * Women with ovulatory factor like PCOS,anovulation and poor ovarian reserve are excluded.
  * Women with endometriosis are excluded.
  * Women with autoimmune diseases like antiphospholipid antibodies or lupus erythematosus are excluded.
  * Documented uterine anomalies, tubal factor, cervical factor and other local causes of infertility.
  * Male factor of infertility is excluded.
  * Bone and metabolic disease, liver diseases and kidney related diseases.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mid aged women with unexplained infertility group and another fertile group to compare vitamin D inbetween them
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2018-01-10 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin D level | 6 months
  Serum vitamin D level in women with unexplained infertility and fertile pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan T Khairy, Professor, Study Director — Hassan tawfek office